IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

## STATISTICAL ANALYSIS PLAN

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment with Desoximetasone 0.25% shampoo (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Scalp Psoriasis

Protocol Number: DSXS1538b Novum Study Number: 71615001

## **Sponsor:**

Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive Hawthorne, NY 10532

## **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

April 24, 2017

Final Version 1.0

IND#124879

Protocol/Study No. DSXS1538b/71615001

Desoximetasone 0.25% Shampoo

# SAP FINAL VERSION APPROVALS

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment with Desoximetasone 0.25% shampoo (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Scalp Psoriasis

| 777 1. TO | |
|---|---|
| Written By: Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 04/24/2017 |
| Reviewed By: Signature: Pina D'Angelo, MSc Senior Director, Scientific Affairs (Biostatistics) Novum Pharmaceutical Research Services | Date: 04/24/2017 |
| Approved By: Signature: James Lee Director, Clinical Research Taro Pharmaceuticals U.S.A., Inc. | Date: 4-24-2017 |

IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|-----------|----------------|--------------------------|-------------|
| Draft 1.0 | April 18, 2017 | New Document | Jianhua Liu |
| Final 1.0 | April 24, 2017 | Finalize SAP | Jianhua Liu |

IND # 124879

Protocol/Study No. DSXS1538b/71615001

Desoximetasone 0.25% Shampoo

# **List of Abbreviations and Definition of Terms**

| Abbreviation | Term |
|--------------|------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| BP | Blood Pressure |
| С | Celsius |
| CRF | Case Report Form |
| CRO | Clinical Research Organization |
| CDISC | Clinical Data Interchange Standards Consortium |
| FDA | Food and Drug Administration |
| HR | Heart Rate |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IGA | Investigator's Global Assessment |
| IND | Investigational New Drug |
| ml | Milliliter |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SDTM | Study Data Tabulation Model |

IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

# **TABLE OF CONTENTS**

| 1. INTRODUCTION | 7 |
|---|---|
| 2. OBJECTIVES | |
| 3. OVERALL STUDY DESIGN | 7 |
| 4. SAMPLE SIZE | |
| 5. STUDY ENDPOINTS AND ANALYSIS POPULATIONS | 10 |
| 6. STATISTICAL ANALYSIS METHODS | 10 |
| 6.1 Baseline Characteristics. | 10 |
| 6.1.1 Demographics | 10 |
| 6.1.2 Medical History | 11 |
| 6.1.3 Physical Exam | |
| 6.1.4 Percent Scalp Affected | 11 |
| 6.1.5 Pregnancy Test | |
| 6.1.6 Concomitant Medications | 12 |
| 6.2 Statistical Analyses | |
| 6.2.1 Safety Analysis of Potential HPA Axis Suppression | |
| 6.2.2 Investigator Global Assessment | |
| 6.3 Safety Analysis | |
| 6.3.1 Adverse Events | |
| 6.3.2 Vital Signs | |
| 6.3.3 Laboratory Evaluation | |
| 6.3.4 Ocular Discomfort Assessment | |
| 6.4 Multiple Comparisons | |
| 6.5 Methods for Handling Missing Data | |
| 6.6 Interim Analyses | 14 |
| 7. TABLE, LISTING AND FIGURE SHELLS | |
| T16.1.9.1 Summary of Patient Disposition | |
| T16.1.9.2 Summary of Protocol Deviations (Safety Population) | |
| T16.1.9.3 Summary of Demographic Data (Safety Population) | |
| T16.1.9.4 Summary of Frequency of HPA Axis Suppression at the End of Treatment | |
| T16.1.9.5 Summary of Percent Scalp Affected with Plaque Psoriasis (Safety Population) | |
| T16.1.9.6 Summary of Frequency of Investigator Global Assessment (IGA) (Safety Popul | |
| T16.1.9.7 Overall Summary of Adverse Events (Safety Population) | 22 |
| T16.1.9.8.1 Summary of Frequency of All Adverse Events by Body System (Safety | 22 |
| Population) | |
| T16.1.9.8.2 Summary of Frequency of All Adverse Events in $\geq 2\%$ of Patients by Body States and States are supported by Events in $\geq 2\%$ of Patients by Body States and States are supported by Events in $\geq 2\%$ of Patients by Body States are supported by Events and Events are supported by Events and Events are supported by Events and Events are supported by Events and Events are supported by Events are supported by Events are supported by Events and Events are supported by Events and Events are supported by Events are supported by Events are supported by Events and Events are supported by Events are supported by Events are supported by Events are supported by Events are supported by Events and Events are supported by Events are sup | |
| (Safety Population) | 23 |
| T16.1.9.10 Summary of Frequency of All Adverse Events by Relationship (Safety Popula | |
| T16.1.9.11 Summary of Frequency of Serious Adverse Events (Safety Population) | 26 |

# IND # 124879

# Protocol/Study No. DSXS1538b/71615001

# Desoximetasone 0.25% Shampoo

| T16.1.9.12 Shift Analysis of Clinical Chemistry Laboratory Results from Bas | eline to End of |
|---|---|
| Treatment (Safety Population) | 27 |
| T16.1.9.13 Shift Analysis of Clinical Hematology Laboratory Results from Ba | aseline to End of |
| Treatment (Safety Population) | |
| L16.2.1 Listing of Discontinued Patients | 28 |
| L16.2.2 Listing of Protocol Deviations | 29 |
| L16.2.3 Listing of Patients Excluded from Safety Analysis of Potential HPA | Axis Suppression30 |
| L16.2.4.1 Listing of Demographic Data | 31 |
| L16.2.4.2 Listing of Medical History | |
| L16.2.4.3 Listing of Concomitant Medication | 33 |
| L16.2.5.1 Listing of Drug Administration. | |
| L16.2.5.2 Listing of Study Medication Weight | |
| L16.2.6.1 Listing of Cortisol Response Test Results | |
| L16.2.6.2 Listing of HPA Axis Suppression Follow-Up | |
| L16.2.6.3 Listing of Investigator Global Assessment (IGA) | |
| L16.2.6.4 Listing of Percent Scalp Affected with Plaque Psoriasis | 39 |
| L16.2.7 Listing of Adverse Events | |
| L16.2.8.1 Listing of Positive Pregnancy Test Results | |
| L16.2.8.2 Listing of Vital Signs | |
| L16.2.8.3 Listing of Abnormal Physical Examination Results | |
| L16.2.8.4 Listing of Clinical Hematology Laboratory Results | |
| L16.2.8.5 Listing of Clinical Chemistry Laboratory Results | |
| L16.2.8.6 Listing of Ocular Signs/Symptoms Assessment | |
| 8. APPENDICES | |
| APPENDIX A: Investigator Global Assessment (IGA) | |
| APPENDIX B: Percent Scalp Affected | |
| APPENDIX C: Ocular Discomfort Assessment | |
| APPENDIX D: Cortisol Response Test | |
| APPENDIX F: Clinical Laboratory Testing | 52 |

IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol DSXS1538b (Study No. 71615001) Rev. 1 dated 06/28/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Clinical Study Protocol DSXS1538b (Study No. 71615001) Rev. 1 dated 06/28/2016
- Case Report Form Booklet Version 1.0 for Study No. 71615001 (DSXS1538b)

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the potential of desoximetasone 0.25% shampoo to suppress HPA axis function in patients with moderate to severe scalp psoriasis.
- 2. Evaluate the efficacy parameters and adverse event (AE) profiles of desoximetasone 0.25% shampoo administered to patients with moderate to severe scalp psoriasis.

## 3. OVERALL STUDY DESIGN

This open-label, safety study is designed to evaluate the potential for adrenal suppression after maximal use treatment with desoximetasone 0.25% shampoo (Taro Pharmaceuticals, U.S.A.), for the treatment of moderate to severe scalp psoriasis.

Up to 5-10 eligible patients with stable plaque psoriasis of the scalp that satisfy all eligibility criteria will be enrolled into the study at Visit 1. Patients must be overall in good health. They should have a current diagnosis of moderate to severe scalp psoriasis with IGA score of at least 3 or 4.

#### IND # 124879

Protocol/Study No. DSXS1538b/71615001

# **Desoximetasone 0.25% Shampoo**

Patients enrolled in the study will apply product once daily for 28 days, according to provided instructions. Each patient is expected to receive 28 doses of study product.

Patients will attend a total of 3 Clinic Visits and a telephone follow-up phone call (Visit 4) as follows:

- Visit 1 (Day 1): Enrollment
- Visit 2 (Day 14±2): Interim Visit
- Visit 3 (Day  $29 \pm 2$ ): End of Study or Early Termination
- Visit 4 (Day 42± 4): Follow-up Telephone Phone Call

The primary endpoint is the proportion of patients in the study with HPA axis suppression following treatment with the study medication.

The safety profile of each treatment group will be evaluated by comparing adverse events.

IND # 124879 Desoximetasone 0.25% Shampoo Protocol/Study No. DSXS1538b/71615001

# **Study Schematic**

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| Day | 1 | 14 ± 2 | 29 ± 2 | 42 ± 4 |
| Procedures | Screening/<br>Enrollment<br>Before 12 pm | Interim<br>Visit | End of<br>Study/Early<br>Termination<br><b>Before 12 pm</b> | Telephone<br>Follow-Up<br>Visit |
| Informed Consent | X | | | |
| Medical History and<br>Demographics | X | | | |
| Vital Signs | X | X | X | |
| Pregnancy Test* | X | X | X | |
| Physical Exam | X | | X | |
| HEENT Exam | X | X | X | |
| % Scalp Affected | X | X | X | |
| Investigator Global Assessment | X | X | X | |
| Concomitant Medication | X | X | X | X |
| Laboratory Evaluations | X | | X | |
| Cortisol Response Test | X | | X | |
| Confirm Inc/Exc Criteria | X | | | |
| Dispense Wristband | X | | | |
| Weigh and Dispense Study Product | X | X | | |
| Collect and Weigh Study Product | | X | X | |
| Dispense/Review Patient Diary | X | X | X | |
| Ocular Assessment | | X | X | |
| Adverse Events | | X | X | X |
| Evaluation of Patient Compliance to the Protocol | | X | X | |

<sup>\*</sup> Pregnancy test will be carried out for females of childbearing potential.

#### IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

#### 4. SAMPLE SIZE

The sample size of 5-10 evaluable patients was deemed appropriate to meet the objective of the study.

#### 5. STUDY ENDPOINTS AND ANALYSIS POPULATIONS

#### **Primary Outcome Measures:**

Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of treatment defined by the following criteria: 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml during the Cortisol Response Test.

The primary endpoint is the proportion of patients in the study with HPA axis suppression following treatment with the study medication.

## **Safety Population:**

Safety Population includes all patients who applied at least one dose of study drug.

#### 6. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include number of observations, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

## **6.1 Baseline Characteristics**

## 6.1.1 Demographics

Demographic information collected at baseline includes the following:

- Age (years)
- Gender (Male/Female)

#### IND # 124879

Protocol/Study No. DSXS1538b/71615001

# **Desoximetasone 0.25% Shampoo**

- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)

Summary tables will be presented. Continuous variables will be summarized using descriptive statistics (n, median, minimum, maximum, mean, standard deviation). Categorical variables will be summarized using frequencies and percentages.

All data will be listed by patient.

## **6.1.2 Medical History**

At Visit 1, patients will be questioned about medical history, including acute and chronic medical history and medical history relevant to their scalp psoriasis.

Medical history data will be listed by patient.

## 6.1.3 Physical Exam

A general physical exam will be conducted at Visit 1 and Visit 3. The physical exam must include a dermatological examination as a minimum.

Abnormal physical exam results will be listed by patient and visit.

## **6.1.4 Percent Scalp Affected**

Patient's scalp will be examined by Investigator/designated clinician to determine the percent surface area affected with plaque psoriasis at all visits.

Descriptive summary (n, mean, standard deviation, median, minimum, maximum) will be presented for percent scalp affected by visit.

Percent scalp affected will be listed by patient and visit.

#### **6.1.5 Pregnancy Test**

Urine pregnancy tests on females of child-bearing potential will be performed at Visit 1, 2 and 3.

Positive pregnancy test results will be listed by patient and visit.

IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

#### 6.1.6 Concomitant Medications

At Visits 1-3 and during the telephone follow-up phone call (Visit 4) patients will be questioned about current and concomitant medication use over the previous 12 weeks. At all Interim Visits patients will be questioned about ongoing or new concomitant medication use.

All prior and concomitant medications taken since screening will be listed by patient.

# **6.2 Statistical Analyses**

## 6.2.1 Safety Analysis of Potential HPA Axis Suppression

Dosing will be once daily for 28 days. Patients who have normal adrenal function at baseline, use at least 21 doses of the study product and have data from a post-treatment cortisol response test will be included in the analysis.

The primary analysis of interest is to assess the proportion of patients considered to have demonstrated possible HPA axis suppression following treatment with the study medication.

A logistic regression of the proportion of patients in the study with HPA axis suppression may be performed as exploratory analysis with % scalp affected as a covariate. This will depend on the distribution of the % scalp data collected. See Appendix D for results from the cortisol response test considered indicative of potential HPA axis suppression.

#### 6.2.2 Investigator Global Assessment

Patient will be examined to determine the severity of scalp psoriasis based on a global assessment of plaque elevation, scaling and erythema by the Investigator/designated clinician.

Investigator Global Assessment data will be summarized using frequency and percentage by visit.

Investigator Global Assessment data will also be listed by patient and visit.

# **6.3 Safety Analysis**

Safety analysis will be conducted on all patients who applied at least one dose of study drug.

#### **6.3.1 Adverse Events**

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities Version 1 or higher) coding dictionary. Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

#### IND # 124879

Protocol/Study No. DSXS1538b/71615001

# **Desoximetasone 0.25% Shampoo**

All AEs will be listed by patient.

A summary table of the number and percent of patients with AEs by system organ class, preferred term will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where "Related includes "Possible", "Probable", or "Definite".

# 6.3.2 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1, 2, and 3.

Vital sign data will be listed by patient and visit.

## **6.3.3** Laboratory Evaluation

At Visit 1 and Visit 3 a blood sample will be collected for hematology and clinical chemistry testing.

Shift analysis using the categories, below, above and within the laboratory normal range will be performed to identify any specific laboratory parameter that shows a trend toward potentially clinically significant changes.

All data will be listed by patient and visit.

## **6.3.4 Ocular Discomfort Assessment**

At Visits 2 and 3 the patient will be asked to assess if any ocular discomfort was experienced, YES or NO, since the last clinic visit. If YES is reported, the patient will be asked to report the signs and symptoms experienced.

All data will be listed by patient and visit.

IND # 124879

Protocol/Study No. DSXS1538b/71615001

**Desoximetasone 0.25% Shampoo** 

## **6.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

# 6.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

# 6.6 Interim Analyses

There is no interim analysis planned in this study.

# 7. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

Novum Pharmaceutical Research Services Protocol/Study No. DSXS1538b/71615001

TABLE, LISTING AND FIGURE SHELLS

**T16.1.9.1 Summary of Patient Disposition** 

| Patients | Total |
|---|---|
| Enrolled | XX |
| Completed Study | XX |
| Terminated Early | XX |
| Adverse event | XX |
| Enrolled in error | XX |
| Lack of efficacy | XX |
| Lost to follow-Up | XX |
| Non-compliance with study drug | XX |
| Non-compliance with study procedure | XX |
| Restricted medication used for the treatment of psoriasis | XX |
| Restricted medication used for reasons other than the treatment of psoriasis | XX |
| Significant worsening of scalp psoriasis required alternative or supplemental therapy | XX |
| Withdrawal by subject | XX |
| Other | XX |

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Total |
|----------------------------------------------------------------------|-------|
| Total Patients with Protocol Deviations | XX |
| Total Deviations | XX |
| Assessment conducted out of window | XX |
| Enrolled in error | XX |
| Lost to follow-up | XX |
| Missed blood collection | XX |
| Missed visit | XX |
| Outside visit window | XX |
| Non-compliance with study drug | XX |
| Non-compliance with study procedure | XX |
| Restricted medication use | XX |
| Study product not applied approximately 24 hours before clinic visit | XX |
| Other | XX |

T16.1.9.3 Summary of Demographic Data (Safety Population)

| | | Total |
|-------------|-------------------------------------------|-----------------|
| | | N=xx |
| Age (years) | n | XX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ |
| | Median | XX.X |
| | Range | xx.x - xx.x |
| Race | American Indian or Alaska Native | xx (xx.x%) |
| | Asian | xx (xx.x%) |
| | Black/African American | xx (xx.x%) |
| | Native Hawaiian or other Pacific Islander | xx (xx.x%) |
| | White | xx (xx.x%) |
| | Other | xx (xx.x%) |
| Ethnicity | Hispanic or Latino | xx (xx.x%) |
| | Not Hispanic or Latino | xx (xx.x%) |
| Gender | Female | xx (xx.x%) |
| | Male | xx (xx.x%) |

N= number of patients; n= number of patients with data available; % is based on N

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Frequency of HPA Axis Suppression at the End of Treatment

| | * * |
|----------------------|------------|
| | Total |
| HPA Axis Suppression | N=xx |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |

N= number of patients included in HPA axis suppression analysis; % is based on N

Created on: ddmmmyy hh:mm


T16.1.9.5 Summary of Percent Scalp Affected with Plaque Psoriasis (Safety Population)

| Visit | n | Mean | SD | Median | Min | Max |
|-------|----|------|------|--------|------|------|
| 1 | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| 2 | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| 3 | xx | XX.X | XX.X | XX.X | XX.X | XX.X |

T16.1.9.6 Summary of Frequency of Investigator Global Assessment (IGA) (Safety Population)

| Visit | 0 (Clear) | 1 (Minimal) | 2 (Mild) | 3 (Moderate) | 4 (Severe) |
|-------|------------|-------------|------------|--------------|------------|
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>%</sup> is based on number of patients included in safety population.

Created on: ddmmmyy hh:mm


T16.1.9.7 Overall Summary of Adverse Events (Safety Population)

| D | Total |
|-----------------------------------------|------------|
| Description | N=xx |
| Patients Randomized | XX |
| Patients with at least one AE | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) |
| AEs reported | XX |
| Mild | xx (xx.x%) |
| Moderate | xx (xx.x%) |
| Severe | xx (xx.x%) |
| Not Related | xx (xx.x%) |
| Related | xx (xx.x%) |
| Death | xx (xx.x%) |
| Serious AE | xx (xx.x%) |

Related = Possible, Probable, Definite

Created on: ddmmmyy hh:mm

T16.1.9.8.1 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| Body System | MedDRA Term | Events | Patients |
|-------------------------------|-------------|--------|------------|
| Patients with at least one AE | Total | XX | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | XX | xx (xx.x%) |

% is based on number of patients included in safety population.

T16.1.9.8.2 Summary of Frequency of All Adverse Events in ≥ 2% of Patients by Body System (Safety Population)

T16.1.9.9 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | , | • • | | |
|---|---|---|---|---|
| Body System | MedDRA Term | Mild | Moderate | Severe |
| Patients with at least one AE | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

% is based on number of patients included in safety population.

T16.1.9.10 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| Body System | MedDRA Term | Related | Not Related |
|-------------------------------|-------------|------------|-------------|
| Patients with at least one AE | Total | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx (xx.x%) | xx (xx.x%) |

Related = Possible, Probable, Definite

Created on: ddmmmyy hh:mm


<sup>%</sup> is based on number of patients included in safety population.

T16.1.9.11 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | MedDRA Term | Total<br>N=xx |
|---|---|---|
| Injury, poisoning and procedural complications | Alcohol poisoning | XX |

Created on: ddmmmyy hh:mm


T16.1.9.12 Shift Analysis of Clinical Chemistry Laboratory Results from Baseline to End of Treatment (Safety Population)

Alanine Aminotransferase (U/L)

| Baseline-> | | | |
|------------|------------|------------|------------|
| Endpoint | Low | Normal | High |
| Low | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| High | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>%</sup> is based on number of patients included in safety population.

Table will continue for other lab parameters.

Similar table will be created for T16.1.9.13.

T16.1.9.13 Shift Analysis of Clinical Hematology Laboratory Results from Baseline to End of Treatment (Safety Population)

**L16.2.1 Listing of Discontinued Patients** 

| Patient<br>Number | Date of<br>Discontinuation | Discontinuation<br>Reason |
|---|---|---|
| XX-XXXX | yyyy-mm-dd | Adverse event |
| XX-XXXX | yyyy-mm-dd | Lost to follow-up |

**L16.2.2** Listing of Protocol Deviations

| Patient<br>Number | Event Description |
|-------------------|--------------------------------|
| XX-XXXX | Outside Visit Window (Visit 3) |

Created on: ddmmmyy hh:mm

# L16.2.3 Listing of Patients Excluded from Safety Analysis of Potential HPA Axis Suppression

| Patient<br>Number | Exclusion Reason |
|-------------------|-----------------------------------------|
| XX-XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Created on: ddmmmyy hh:mm


L16.2.4.1 Listing of Demographic Data

| Patient<br>Number | Age | Gender | Ethnicity | Race |
|---|---|---|---|---|
| XX-XXXX | 30 | Female | Not Hispanic or Latino | Black or African American |

# L16.2.4.2 Listing of Medical History

| Patient<br>Number | System | Diagnosis or<br>Surgical Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|
| XX-XXXX | Gynecologic | Menopause | yyyy-mm-dd | yyyy-mm-dd | |

Created on: ddmmmyy hh:mm


# L16.2.4.3 Listing of Concomitant Medication

| Patient<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Location | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| XX-XXXX | No | Advil | 2 TAB | QD | Oral | XXXXXXXX | yyyy-mm-dd /<br>yyyy-mm-dd | Cold |

# L16.2.5.1 Listing of Drug Administration

| Patient | Date of | Date of | Total | Compliance |
|---------|------------|------------|---------------|------------|
| Number | First Dose | Last Dose | Doses Applied | (%) |
| xx-xxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX.X |

#### Note to programmer:

Compliance = [Total number of applications] / [Planned number of applications] \* 100%, where Planned number of applications is determined as follows: for subjects who completed the study successfully: 28 applications (28 days of once daily dosing);

for subjects who discontinued early: the minimum between 28 and [(Date of Discontinuation – Date of First Application)+1].

Created on: ddmmmyy hh:mm


L16.2.5.2 Listing of Study Medication Weight

| Patient — Number | Bottle 1 | | Bottle | Total | |
|---|---|---|---|---|---|
| | Weight<br>Dispensed | Weight<br>Collected | Weight<br>Dispensed | Weight<br>Collected | Amount<br>Applied |
| | (g) | (g) | (g) | (g) | (g) |
| XX-XXXX | XX | XX | XX | XX | XXX |

L16.2.6.1 Listing of Cortisol Response Test Results

| ' | | | | | | | Basal | Post Injection | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Was a Cortisol | | | | Post- | Cortisol | Cortisol | Have | |
| Patient<br>Number V | | Response Test conducted? | Date I | Basal Sample<br>Draw Time | Injection<br>Time | Injection | Concentration | Concentration | Abnormal | |
| | Visit | | | | | Draw | Level | Level | Adrenal | HPA axis |
| | | | | | | Time | (mcg/100ml) | (mcg/100ml) | Function? | Suppression |
| XX-XXXX | 1 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | No | No |
| | 3 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | Yes | No |
| XX-XXXX | 1 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | No | No |
| | 3 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | Yes | Yes |
# L16.2.6.2 Listing of HPA Axis Suppression Follow-Up

| | | | _ | | _ | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Number | Is The Patient Showing Signs<br>Or Symptoms Of HPA Axis<br>Suppression?/<br>Was a Cortisol Response<br>Test Conducted? | Follow-Up<br>Test | Date/ Basal Sample Draw Time/ Injection Time/ Post-Injection Draw Time | Basal<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Post Injection Cortisol Concentration Level (mcg/100ml) | Still Show<br>Signs of<br>HPA Axis<br>Suppression? | Was the Patient Referred to an Endocrinologist |
| | | | yyyy-mm-dd / hh:mm / | XXX | XXX | No | No |
| XX-XXXX | Yes/ Yes | Test 1 | hh:mm/ hh:mm | | | | |

L16.2.6.3 Listing of Investigator Global Assessment (IGA)

| Patient<br>Number | Visit 1 | Visit 2 | Visit 3 / Early<br>Termination |
|-------------------|---------|---------|--------------------------------|
| XX-XXXX | 0 | 0 | 0 |

### L16.2.6.4 Listing of Percent Scalp Affected with Plaque Psoriasis

| Patient<br>Number | Visit 1 | Visit 2 | Visit 3 / Early<br>Termination |
|-------------------|---------|---------|--------------------------------|
| XX-XXXX | XXX | XXX | XXX |

Created on: ddmmmyy hh:mm

# **L16.2.7 Listing of Adverse Events**

| Patient<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment<br>Area | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action Taken | SAE? |
|---|---|---|---|---|---|---|---|---|
| xx-xxxx | Nervous system disorders / | No | yyyy-mm-dd / | Mild | Not Related | Recovered | Dose Not Changed/ | No |
| | Headache / | | yyyy-mm-dd | | | | None | |
| | Headache | | | | | | | |

L16.2.8.1 Listing of Positive Pregnancy Test Results

| Patient<br>Number | Visit 1 | Visit 2 | Visit 3 |
|-------------------|----------|----------|----------|
| xx-xxxx | Negative | Negative | Positive |

L16.2.8.2 Listing of Vital Signs

| Patient<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP (mmHg) | Heart Rate (beats/min) | Respiration Rate (breaths/min) | Temperature (F) |
|---|---|---|---|---|---|---|
| xx-xxxx | 1 | 120 | 70 | 84 | 18 | 98.6 |
| | 2 | 140 | 80 | 74 | 18 | 97 |
| | 3 | 130 | 87 | 74 | 18 | 99.2 |

L16.2.8.3 Listing of Abnormal Physical Examination Results

| - : | | | |
|---------|--------|--------|-----------------|
| Patient | Visit | System | Results |
| Number | V 1510 | System | resures |
| XX-XXXX | 1 | HEENT | Abnormal (Scar) |
| | 2 | | |
| | 3 | | |

L16.2.8.4 Listing of Clinical Hematology Laboratory Results

| | | _ | | | ~ | |
|---|---|---|---|---|---|---|
| Patient<br>Number | Visit | Hematocrit (L/L) | Basophils (10^9/L) | Platelets (10^9/L) | Hemoglobin (g/L) | etc. |
| XX-XXXX | 1 | XXX | XXX | XXX | XXX | XXX |
| | 3 | XXX | XXX | XXX | xxx (Low) | XXX |

L16.2.8.5 Listing of Clinical Chemistry Laboratory Results

| Patient<br>Number | Visit | Alkaline<br>Phosphatase<br>(U/L) | Alanine<br>Transaminase<br>(U/L) | Aspartate<br>Transaminase<br>(U/L) | Blood Urea<br>Nitrogen<br>(mmol/L) | etc. |
|---|---|---|---|---|---|---|
| XX-XXXX | 1 | XXX | XXX | xxx (High) | XXX | XXX |
| | 3 | XXX | XXX | XXX | XXX | XXX |

# L16.2.8.6 Listing of Ocular Signs/Symptoms Assessment

| Patient<br>Number | Visit | Did the patient experience any ocular discomfort? | Signs/Symptoms the patient experienced | Did the shampoo come into contact with the patient's eyes? | Patient's overall discomfort |
|---|---|---|---|---|---|
| XX-XXXX | 2 | Yes | Redness/Pain | Yes | Mild |
| | 3 | No | | | |
| XX-XXXX | 2 | Yes | Itching/Pain | Yes | None |
| | 3 | Yes | Itching/Pain | No | |

### 8. APPENDICES

# **APPENDIX A: Investigator Global Assessment (IGA)**

To be eligible for inclusion in the study the IGA must be 3 or 4 at baseline. Patients will be considered to have shown improvement in disease severity if the IGA score decreases by at least one unit from the baseline score, and will be considered a treatment success if the IGA score decreases at least 2 units from the baseline score.

| Score | Category | Description |
|---|---|---|
| 0 | Clear | Plaque elevation: no evidence of plaque elevation above normal skin level Scaling: no evidence of scaling |
| | | Erythema: no redness |
| 1 | Minimal | Plaque elevation: very slight elevation above normal skin level, easier felt than seen |
| | | Scaling: limited amount of very fine scales partially covers some of the plaques |
| | | Erythema: very few of the plaques are light red |
| 2 | Mild | Plaque elevation: slight but definite elevation above the normal skin level, typically with edges that are indistinct or sloped on some of the plaques |
| | | Scaling: mainly fine scales, some plaques are partially covered Erythema: some plaques are light red |
| 3 | Moderate | Plaque elevation: moderate elevation with rounded or sloped edges on most of the plaques |
| | | Scaling: somewhat coarser scales; most plaques are partially covered |
| | | Erythema: most plaques are red |
| 4 | Severe | Plaque elevation: marked to very marked elevation, with hard to very hard sharp edges on virtually all or all of the plaques |
| | | Scaling: coarse, thick scales; virtually all or all plaques are covered; rough surface |
| | | Erythema: virtually all or all plaques are bright to dusky red |

### **APPENDIX B: Percent Scalp Affected**

Investigators will use the following chart to identify areas and estimate scalp surface area affected by psoriasis plaques. <sup>16</sup>



Olsen/Canfield

### **APPENDIX C: Ocular Discomfort Assessment**

At Visits 2 and 3 the patient will be asked to assess if any ocular discomfort was experienced, YES or NO, since the last clinic visit.

If YES is reported, the patient will be asked to report the signs and symptoms that apply from the list below or indicate any OTHER signs and symptoms experienced:

Redness Stinging

Itching Blur (decrease in vision)

Pain Increased sensitivity

Swelling Watery eyes

Burning Spots, flashes and floaters

Eye Discharge Foreign body sensation

In addition, the patient will be asked to indicate if the shampoo came into contact with their eye, YES or NO, since the last clinic visit. If YES is reported, the patient will be asked to rate the discomfort at the time of contact as None, Mild, Moderate or Severe.

### **APPENDIX D: Cortisol Response Test**

This cortisol release test is modified from the procedure of Wood et al as described in the Product Label for Cortrosyn<sup>TM</sup> (cosyntropin) for injection (Amphstar Pharmaceuticals, Inc.).

The procedure is as follows:

- 1. A single 5 ml blood sample should be taken as the basal sample.
- 2. 0.25 mg (a single vial) of Cortrosyn<sup>TM</sup> (cosyntropin) should be reconstituted with 1.0ml of 0.9% sodium chloride injection USP injected intramuscularly. In patients under 3 years of age, 0.125mg of Cortrosyn<sup>TM</sup> will be used.
- 3. 30 minutes after the IM injection a second 5 ml blood sample should be obtained. The resulting two serum samples (at least 1 ml of serum in each) should be processed and labeled according to the instructions provided and sent the same day to ACM Global Laboratory for analysis of basal and post stimulated serum cortisol concentration.

The resulting blood samples should be sent to ACM Global Laboratory for immediate testing.

The test at the End of Study visit should not be performed if the patient dosed within 12 hours.

A patient will be considered to have normal basal cortisol level and adrenal function if they meet all three criteria listed below under Normal. Failure to meet any of these criteria is indicative of abnormal adrenal function or potential HPA axis suppression.

| | Cortisol Results | |
|---|---|---|
| | Normal | Abnormal |
| Basal (pre Cortrosyn <sup>TM</sup> injection) | ≥ 5 mcg/100ml | < 5 mcg/100ml |
| 30 minutes post | ≥ basal value + 7 | < basal value + 7 |
| Cortrosyn <sup>TM</sup> injection | > 18 mcg/100ml | ≤ 18 mcg/100ml |

HPA Axis suppression will be defined as a 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml. If the Visit 1 Cortisol Response Test shows signs of HPA axis suppression as defined above the patient will be contacted and instructed to discontinue the use of study product, not to iniate any new steroid therapy, topical or otherwise and an End of Study Visit will be scheduled to conduct a Cortisol Response Test at least 28 days after the initial Cortisol Response Test at Visit 1 to assess for HPA axis suppression. At Visit 3 the study treatment period will be over, any patients with results of HPA axis suppression will be advised not to initiate any new steroid therapy, topical or otherwise, and to return to the site in 28 days at which time they will be assessed for HPA axis suppression.

Any patient presenting with symptoms of HPA axis suppression, such as nausea, headache, myalgia, fatigue or loose stool, will be referred to an endocrinologist. As an

additional safety precaution, wristbands identifying the patient as someone suffering from adrenal suppression secondary to steroid withdrawal will be provided to alert medical personnel should any emergencies arise before adrenal function returns to normal.

If the results of the cortisol response test still show signs of HPA axis suppression 28 days after discontinuing therapy they will be asked to return in 28 days (56 days after discontinuing steroid therapy) for another follow-up test. If the patient is still showing signs of HPA axis suppression 56 days after discontinuing steroid therapy and presents with related symptoms they will be referred to an endocrinologist.

If HPA axis suppression persists for 56 days after discontinuing steroid therapy, but the patient has no symptoms they will be asked to return in 28 days (84 days after discontinuing steroid therapy) for another follow-up test. If HPA axis suppression persists for 84 days after discontinuing steroid therapy patients will be referred to an endocrinologist regardless of symptoms.

Patients should not be subjected to Cortrosyn<sup>TM</sup> testing, or any other challenge to their adrenal response, any sooner than 4 weeks from their last Cortrosyn<sup>TM</sup> test.

Follow-Up Schedule for Patients showing signs of HPA Axis Suppression

| Days<br>after d/c | HPA Results | Symptom s | Patient Course |
|-------------------|-------------|-----------|-----------------------------|
| 28 | Normal | N/A | Study over |
| 28 | Abnormal | Yes | Refer to endocrinologist |
| 28 | Abnormal | No | Repeat test in 28 days |
| 56 | Normal | N/A | Study over |
| 56 | Abnormal | Yes | Refer to endocrinologist |
| 56 | Abnormal | No | Repeat test in 28 days |
| 84 | Normal | N/A | Study over |
| 84 | Abnormal | Yes or No | Refer to an endocrinologist |

### **APPENDIX F: Clinical Laboratory Testing**

As part of the Screening Procedures and at Visit 3 (or early termination for randomized patients only) patients will have a blood sample taken for hematology and clinical chemistry testing. The testing panel should include as a minimum the following tests:

#### Hematology

- Hematocrit
- White blood cell count
- Platelets
- Hemoglobin
- Red blood cell count
- Differential white cell count

### Chemistry

- Alkaline phosphatase
- Total bilirubin
- Alanine transaminase
- Creatinine
- Aspartate transaminase
- Glucose
- Blood urea nitrogen

Clinical Laboratory Testing will be performed at a Central Laboratory

#### ACM Medical Lab, Inc.

160 Elmgrove Park

Rochester, NY 14624, USA